CLINICAL TRIAL: NCT02168530
Title: A Study of Oral Vismodegib for the Treatment of Idiopathic Pulmonary Fibrosis (IPF)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB29298; 2014-000963-42 (EudraCT Number)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Vismodegib (Experimental)
  Interventions: Drug: vismodegib

INTERVENTIONS:
Drug: placebo — matching placebo administered daily orally
  Arms: Placebo
Drug: vismodegib — vismodegib 150 mg administered daily orally
  Arms: Vismodegib

SUMMARY:
This is a randomized, multicenter, double-blind, placebo-controlled, parallel-group study of vismodegib in patients with IPF. Eligible patients will be randomized in a 2:1 ratio to one of two treatment arms: vismodegib or placebo. The duration of treatment will be 52 weeks. Study drug will be administered daily by the oral route. An 8-week safety follow-up period is included for all patients who receive at least one dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged >/=40 years at Visit 1
* Diagnosis of IPF within the previous 5 years from time of screening and confirmed at baseline
* Patients from countries where a treatment is licensed/approved for IPF must additionally meet at least one of the following criteria to be eligible: (1) be unable to access a licensed therapy for IPF; (2) treatment with a licensed therapy/therapies has been stopped for lack of efficacy or because of safety/tolerability reasons (a washout period will be required); (3) be unwilling to be treated with a licensed therapy and study enrollment considered appropriate.
* Forced vital capacity (FVC) >/=40% and </=90% of predicted at screening
* Stable baseline lung function as evidenced by a difference of <10% in absolute FVC measurements (in liters) between screening and Day 1/Visit 2 prior to randomization
* Diffusion capacity of the lung for carbon dioxide (DLCO) >/=25% of predicted at screening
* Adequate hematopoietic capacity, liver and renal function
* Female patients of childbearing potential must use two methods of acceptable contraception, including one highly effective method and a barrier method, during treatment and for 7 months after completion of study treatment (or as per local requirement)
* Male patients must agree to remain abstinent or use a condom, even after a vasectomy, during sexual intercourse with female partners while being treated with vismodegib/placebo, and for 2 months after completion of study treatment
* Agreement not to donate blood or blood products during the study and for at least 7 months (or as per local requirements) after the last dose of study treatment

Exclusion Criteria:

* Pregnant or lactating
* Known hypersensitivity to any of the study drug excipients or the drug itself
* Prior treatment with vismodegib or any Hh-pathway inhibitor
* Evidence of other known causes of interstitial lung disease
* Hospitalization due to an exacerbation of IPF within 4 weeks prior to, or during, screening
* Lung transplant expected within 12 months of screening
* Evidence of clinically significant lung disease other than IPF
* Substantial emphysema on high resolution computed tomography (HRCT) with degree of emphysema greater than fibrosis
* Post bronchodilator forced expiratory volume in 1 second/FVC ratio <0.7 at screening
* Class IV New York Heart Association chronic heart failure or historical evidence of left ventricular ejection fraction <35%
* Known current malignancy or current evaluation for a potential malignancy
* Known immunodeficiency, including but not limited to HIV infection
* Any clinically significant medical disease (other than IPF) that is associated with an expected survival of <12 months, likely to require a change in therapy during the study, or likely to impact the ability of the patient to participate in the study in the opinion of the investigator, or impact the study efficacy or safety assessments

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in forced vital capacity (FVC) percent predicted | From baseline to Week 52

SECONDARY OUTCOMES:
Change in diffusion capacity of the lung for carbon dioxide (DLCO) | From baseline to Week 52
Annualized rate of change in FVC | Week 52
Progression-free survival | Week 52
Time from randomization to first event of acute IPF exacerbation | Up to 52 weeks
Change in Quality of Life measurements | From baseline to Week 52
Safety: Incidence of adverse events (AEs) | Approximately 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche